CLINICAL TRIAL: NCT05827705
Title: The Effects of Position and Predictive Factors on Hypotension in Patients Undergoing Prone Percutaneous Nephrolithotomy
Brief Title: Position and Predictive Factors of Hypotension in Prone Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyda Efsun Ozgunay, Asocc Prof, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/03-14
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hypotension; Urolithiasis
Keywords: Hypotension; prone position; nephrolithotomy
MeSH Terms: conditions — Hypotension; Urolithiasis | interventions — Health Services Needs and Demand; Ephedrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group H: General anaesthesia was induced by Propofol (2 mg/kg) IV, Rocuronium (0.6 mg/kg) and Fentanyl (2 μg/kg) IV, and maintained with sevoflurane and Epidural anesthesia, intraoperative Hypotensive patients
  Interventions: Other: need for Ephedrine hydrochloride
- Group N: General anaesthesia was induced by Propofol (2 mg/kg) IV, Rocuronium (0.6 mg/kg) and Fentanyl (2 μg/kg) IV, and maintained with sevoflurane and Epidural anesthesia, intraoperative Non-Hypotensive patients

INTERVENTIONS:
Other: need for Ephedrine hydrochloride — ephedrine dose in hypotension
  Other Names: Need for ephedrine hidroclorur
  Groups: Group H

SUMMARY:
This study was designed to investigate the effect of position and predictive factors on hypotension in patients performing percutaneous nephrolithotomy. Patients aged >18 years and ASA I-III who underwent general or regional anaesthesia were included in the study. Percutaneous access was performed in all patients with fluoroscopy in the prone position.

DETAILED DESCRIPTION:
This study was designed to investigate the effect of position and predictive factors on hypotension in patients performing percutaneous nephrolithotomy. Patients aged >18 years and ASA I-III who underwent general or regional anaesthesia were included in the study. Percutaneous access was performed in all patients with fluoroscopy in the prone position. Age, gender, body mass index(BMI), smoking, type of anaesthesia, duration of anaesthesia and surgery were recorded.

The ECG, SpO2, and non-invasive blood pressure values were recorded intraoperatively. Preoperative and postoperative 12th hour Hb,BUN, Cr,Na,K and Cl were measured in a blood sample. Isotonic was used as an intravenous fluid in all participants. In treatment of hypotension routine ephedrine treatments were recorded.

In the literature, studies in PCNL surgery have focused on data such as method, duration of bleeding and fluoroscopy, electrolyte-metabolic changes, and complications such as fever, hypothermia, pleural damage, and hospital stay. A limited number of studies have focused on bleeding and hemodynamics in comparing surgical methods in the prone and supine positions. the investigators could not find any study comparing systemic disease effects on intraoperative hypotension (hemodynamic parameters) in Prone PCNL surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years and ASA I -III who underwent general or regional anaesthesia were included in the study.

Exclusion Criteria:

* Patients who received preoperative vasopressor, inotropic infusion, erythrocyte and fresh frozen plasma (FFP), anaemia, uncontrolled coagulopathies, pregnancy, immunodeficiency, ASA class IV and emergency surgeries.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients aged >18 years
Study Population: Percutaneous access was performed in all patients with fluoroscopy in the prone position after the ureteral catheter placement in the lithotomy position as standard.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
1.Perioperatif hypotension and presence of systemic diseases | Perioperative period
  Systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <65 mmHg, or a decrease of more than 20% of baseline
Prone position effects on hypotension | Perioperative period
  Systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <65 mmHg, or a decrease of more than 20% of baseline

SECONDARY OUTCOMES:
mortality | 30 days after the surgery
  death

CONTACTS AND LOCATIONS:
Overall Officials: Seyda E Ozgunay, 1, Principal Investigator — Bursa Yüksek İhtisas EAH
Locations (1):
- Bursa yüksek ihtisas EAH, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocal can be shared.
Supporting Information: Study Protocol
Time Frame: One year
Access Criteria: Study Protocol

REFERENCES:
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Vernooij LM, van Klei WA, Machina M, Pasma W, Beattie WS, Peelen LM. Different methods of modelling intraoperative hypotension and their association with postoperative complications in patients undergoing non-cardiac surgery. Br J Anaesth. 2018 May;120(5):1080-1089. doi: 10.1016/j.bja.2018.01.033. Epub 2018 Mar 21. PMID 29661385
- [Background] Melo PAS, Vicentini FC, Perrella R, Murta CB, Claro JFA. Comparative study of percutaneous nephrolithotomy performed in the traditional prone position and in three different supine positions. Int Braz J Urol. 2019 Jan-Feb;45(1):108-117. doi: 10.1590/S1677-5538.IBJU.2018.0191. PMID 30521168
- [Result] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768